CLINICAL TRIAL: NCT03968081
Title: Exploration of Theory of Mind in a Situation of Social Rejection in Borderline Personality Disorder
Acronym: LIMITOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: human ressources
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Paul ROUX, Principal Investigator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P18/12_LIMITOM
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Borderline Personality Disorder; Social Rejection; Social Skills; Cognitive Function 1, Social
Keywords: theory of mind; mentalisation; ostracism; cyberball
MeSH Terms: conditions — Borderline Personality Disorder; Social Isolation; Social Skills; Ostracism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social exclusion (Experimental): Participating at the cyberball game in exclusion condition in wich they will receive 2 time the ball in the 10 first throw then none of them in the last 20 throw.
  Interventions: Behavioral: Cyberball
- Social inclusion (Active Comparator): Participating at the cyberball game in inclusion condition in wich they will receive 33% of the throw : 10 in a total of 30
  Interventions: Behavioral: Cyberball

INTERVENTIONS:
Behavioral: Cyberball — a ball tossing playing game in which the experimentor can control the number of throws received by the participants

SUMMARY:
Theory of mind is one of the features of mentalization. It can be defined as the ability to predict or explain other's behavior with the assignment of beliefs, wishes, and intentions and knowing how to discriminate them with our own, or in other words to know how other people think.

Although this ability is crucial to behave adequately in a complex environment, theory of mind judgments are not always optimal.

Notably, individuals with borderline personality disorder are may have difficulties to infer other people's thought and state of mind as well as their own mental states.

These aspects could be at the origin of symptoms like impaired and unstable relationships, identity disruption and excessive fear of abandonment.

Clinical and scientific point suggest that this struggle can be reinforced by social exclusion.

Our study aims at identifying if a situation of social exclusion (compared with social inclusion) may decrease theory of mind performance in borderline personality disorder.

Participants will play a virtual ball-tossing game on a computer, which can lead to a situation of social inclusion or exclusion. Before and after that, they will perform theory of mind tests with visual material.

The study will address three research questions:

Q1: Is theory of mind performance lowered after social exclusion, compared with social inclusion?

Q2: is the self-reported mentalization skills correlated with theory of mind performances?

Q3: Is the social rejection sensitivity correlated with the the theory of mind performances ?

The investigators make several hypotheses related to the previous research questions:

Q1: the investigators expect social exclusion will decrease the subject's theory of mind performances.

Q2: the investigators expect low mentalization skills are correlated to low theory of mind performances.

Q3: the investigators expect that a high social rejection sensitivity will be correlated with low theory of mind performances.

DETAILED DESCRIPTION:
SAMPLING PLAN

Existing data registration before the creation of data:

As of the date of submission of this research plan for preregistration, the data have not yet been collected, created, or realized.

Data collection procedures. Individuals with a borderline personality disorder will be recruited from community mental health centers. All participants will be naive to the purpose of the study, give informed consent in accordance with institutional guidelines and the Declaration of Helsinki.

Sample size Maximum of 50 individuals with a borderline personality disorder. Given that psychometric properties of intention attribution measures by the VLIS in borderline personality disorder aren't known and the impact of social exclusion lead by a virtual ball-tossing game in intention's attribution aren't know either, it is impossible to operate a calculation of the number of necessary subjects.

However, a previous study has shown that is was possible to prove a significant diminution of theory of mind measure in a group of 17 subjects with a borderline personality disorder, after being socially excluded by the cyberball.

Because the measures used in this study are different from ours, the investigators offer to proceed with an intermediate analysis of power after including 10 subjects in each condition (social exclusion and inclusion).

This power analysis aims to calculate the number of subjects the investigators should recruit for the difference underlined by our two intermediate samples to become significant.

If this number exceeds 25 subjects in each group, the research will be stopped.

DESIGN PLAN

First, the investigators will collect socio-demographic data then the participants will have various evaluations and tests like the MADRS depression scale, the WAIS-IV with matrix reasoning, vocabulary and letter-number sequencing, an executive functions test (Test des commissions).

Before playing the cyberball game the participants will perform the first sequence of intentional cartoon task, a computer task in which the subject had to choose a logical end at a 3 boxes comic strip, involving or not a human intention.

Then they will play the cyberball game, a virtual ball-tossing game in which they are lead to think they are playing online with two other people while it is actually a randomized pre register condition.

Following the VLIS, a theory of mind test in which the subject as to infer intentionality likehood for characters in various movies extracts.

Then the second sequence of intentional cartoon task.

They will finish with the the height items reflexive questionnaire and the VSISR (Versailles Sensitivity for Social Rejection, measuring social rejection sensitivity).

ANALYSIS PLAN

Comparison between groups :

The groups' socio-demographic (age, sex, education), cognitive ( current IQ, and executive performance with planning and working memory) and mood (depression) characteristics will be compared using the Student t test or Χ² tests when appropriate. Only variables that significantly differ between the two groups will be included as covariates in the following analyses.

The first analysis of covariance with repeated measures will be run with VLIS score as the dependent variable, the condition (social exclusion or inclusion) as the independent factor, and depression scale, and cognitive performances (matrix reasoning, vocabulary, letter-number sequencing, and executive functions test) as covariates.

A second analysis of covariance with repeated measures will be run with intentional cartoon task score as the dependent variable, the condition (social exclusion or inclusion) as the independent between-subject factor, the time of measurement (before or after the cyberball) and the cartoon condition (intentional or non intentional) as the independent within-subject factors, and depression scale and cognitive performances (matrix reasoning, vocabulary, letter-number sequencing and executive functions test) as covariates.

The third analysis of covariance with repeated measures will be run with questionnaire of reflexive functions score as the dependent variable, the condition (social exclusion or inclusion) as the independent factor and depression scale, and cognitive performances (matrix reasoning, vocabulary, letter-number sequencing, and executive functions test) as covariables

Correlation analyses

Spearman's correlation will be computed between:

* change in intentional cartoon task score after social exclusion and VSISR
* intentional cartoon task score and questionnaire of reflexive functions score
* VLIS score and questionnaire of reflexive functions score

Missing data management :

The investigators predict an anecdotal quantity of missing data (<5%) in our study. If need be the investigators will exclude them.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V criteria for borderline personality disorder (Structured Clinical Interview for Disorders)

Exclusion Criteria:

* Criteria of DSM-V substance use disorder from moderate to severe (except for tobacco and caffeine) in the last six months
* schizophrenic disorder
* Bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Theory of mind performance | One measure per subject, assessed during a 30 min long task
  Total score at the VLIS (Versailles intentional reading in situation), minimum 0, maximum 90, a low outcome indicate high theory of mind performances whereas a high score indicate low theory of mind performances.
  Accuracy and reaction time at the intentional cartoon task
Evolution of theory of mind performance after cyberball - accuracy | 56 repeated measures per subject, assessed during a 10 min long task
  Accuracy (percentage minium 0 maximum 100) in the intentional cartoon task : a computer task in wich the subjects have to choose the logical end of comic strip involving or not human intention. There is 28 comic strip in each of the two sessions.
Evolution of theory of mind performance after cyberball - reaction time | 56 repeated measures per subject, assessed during a 10 min long task
  Reaction time (milliseconds, minimum 100 milliseconds maximum 4000 milliseconds) in the intentional cartoon task : a computer task in wich the subjects have to choose the logical end of comic strip involving or not human intention. There is 28 comic strip in each of the two sessions.

SECONDARY OUTCOMES:
Mentalization performance | One measure per subject, assessed during a 5 min long interview
  Total score on the 8 item reflexive questionary, a self report scale with 8 items (minimum 0, maximum 56) which measure the subject's mentalization abilities.
  A low outcome reflects low self evaluation of mentalizing skill, whereas a high outcome reflects high self evaluation of mentalizing skills.
Social rejection sensibility - intentional rejection | One measures per subject, assessed during a 20 min long interview
  Using the VSISR which is a self-report scale including 20 items of intentional rejection and 20 match items of non intentional rejection, the subject will rate each one from 0 to 10 as a function of the anticipated suffering (0 for none, 10 for maximum suffering).
  The investigators will use intentional rejection score (minium 0 maximum 200).
Social rejection sensibility - difference between intentional and non intentional rejection | One measures per subject, assessed during a 20 min long interview
  Using the VSISR which is a self-report scale including 20 items of intentional rejection and 20 match items of non intentional rejection, the subject will rate each one from 0 to 10 as a function of the anticipated suffering (0 for none, 10 for maximum suffering).
  The investigators will use difference between intentional and non intentional rejection score (minium 0 maximum 200).

CONTACTS AND LOCATIONS:
Overall Officials: Paul ROUX, MD PHD, Principal Investigator — Versailles Hospital
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savage M, Lenzenweger MF. The Impact of Social Exclusion on "Reading the Mind in the Eyes" Performance in Relation to Borderline Personality Disorder Features. J Pers Disord. 2018 Feb;32(1):109-130. doi: 10.1521/pedi_2017_31_293. Epub 2017 May 17. PMID 28513343
- [Background] Nemeth N, Matrai P, Hegyi P, Czeh B, Czopf L, Hussain A, Pammer J, Szabo I, Solymar M, Kiss L, Hartmann P, Szilagyi AL, Kiss Z, Simon M. Theory of mind disturbances in borderline personality disorder: A meta-analysis. Psychiatry Res. 2018 Dec;270:143-153. doi: 10.1016/j.psychres.2018.08.049. Epub 2018 Sep 21. PMID 30248485
- [Background] Williams KD, Jarvis B. Cyberball: a program for use in research on interpersonal ostracism and acceptance. Behav Res Methods. 2006 Feb;38(1):174-80. doi: 10.3758/bf03192765. PMID 16817529
- [Background] Fonagy P, Bateman A. The development of borderline personality disorder--a mentalizing model. J Pers Disord. 2008 Feb;22(1):4-21. doi: 10.1521/pedi.2008.22.1.4. PMID 18312120
- [Background] Staebler K, Renneberg B, Stopsack M, Fiedler P, Weiler M, Roepke S. Facial emotional expression in reaction to social exclusion in borderline personality disorder. Psychol Med. 2011 Sep;41(9):1929-38. doi: 10.1017/S0033291711000080. Epub 2011 Feb 9. PMID 21306661
- [Background] Bazin N, Brunet-Gouet E, Bourdet C, Kayser N, Falissard B, Hardy-Bayle MC, Passerieux C. Quantitative assessment of attribution of intentions to others in schizophrenia using an ecological video-based task: a comparison with manic and depressed patients. Psychiatry Res. 2009 May 15;167(1-2):28-35. doi: 10.1016/j.psychres.2007.12.010. Epub 2009 Apr 5. PMID 19346006
- [Background] Roux P, Brunet-Gouet E, Passerieux C, Ramus F. Eye-tracking reveals a slowdown of social context processing during intention attribution in patients with schizophrenia. J Psychiatry Neurosci. 2016 Mar;41(2):E13-21. doi: 10.1503/jpn.150045. PMID 26836621